CLINICAL TRIAL: NCT01392729
Title: An Open Label, Prospective, Observational, Local, Non-interventional Study of BeVacizumab (Avastin) and IntErpherone (IFN) Alpha 2a in Patients With Metastatic and Locally Advanced Renal Cell CAncer (VERA Study)
Brief Title: An Observational Study of Avastin (Bevacizumab) and Interferon Alpha 2a in Patients With Metastatic Renal Cell Cancer (VERA)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25255
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective observational study will evaluate the efficacy and safety of Avastin (bevacizumab) in combination with interferon alpha 2a in patients with previously untreated metastatic renal cell cancer. Data will be collected from each patient for up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Histologically confirmed metastatic renal cell cancer, clear cell type
* Eligible for treatment with Avastin and interferon alpha 2a according to local prescribing information

Exclusion Criteria:

* Contraindications for Avastin or interferon alpha 2a treatment according to local Summary of Product Characteristics
* Known hypersensitivity to Avastin and/or interferon alpha 2a or any of its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with previously untreated metastatic renal cell cancer
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | approximately 4 years

SECONDARY OUTCOMES:
Overall survival | approximately 4 years
Response rate | approximately 4 years
Safety: Incidence of adverse events | approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Cluj-Napoca, Romania